CLINICAL TRIAL: NCT03185273
Title: In-depth Exploration of a Bidirectional Parent-child Relationship and Its Mediating and Moderating Factors Among Low-income Families in Hong Kong
Brief Title: Parent-child Relationship Among Low-income Families in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW16-145
Record Dates: First submitted 2017-05-25; First posted 2017-06-14 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Child Development; Parent-Child Relations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from buccal epithelial cells. Telomere length will be measured by the method adapted from that originally published by Cawthon. For each sample, the telomere length will be represented by the relative ratio of the telomere repeat copy number (T) to the single copy gene 36BA copy number (S). The T/S ratio will be determined by quantitative polymerase chain reaction (qPcR) using a 7900HT Thermocycler (Applied Biosystems).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective cohort study building upon the existing cohort study on the effectiveness of the Trekkers Family Enhancement Scheme. This study will sample 200 low-income parent-child pairs and follow them up for 24 months with yearly assessment on parental stress and child health using both subjective measures and objective physiological parameters. Additional data on parenting style, neighbourhood cohesion, child physical assault and neglect potential, parental mental health and HRQOL and family disharmony will also be collected at each assessment time point for testing mediating and moderating mechanisms between parental stress and child health. The baseline assessment will be carried out in 2016-17 with three repeated assessments after 6 months, 12 months, and 24 months.

DETAILED DESCRIPTION:
Study aims

* To examine the relationship between parental stress and child health.
* To evaluate the stress of parents as indicated by their subjective perception of mental health, quality of life and allostatic load on the body.
* To evaluate the health of children as indicated by their well-being, behaviors, body mass index (BMI) z-score and telomere length.
* To examine the correlation between changes in parental stress and changes in child health over time.
* To identify the moderators and mediators of the relationship between parental stress and child health.

Eligible participants in the main cohort study will be approached by call or during face-to-face sessions. Parents who express interest in participation will be provided with an information sheet about the research and asked to sign the consent form for themselves and for their children. After providing consent, the parent of each parent-child pair will complete a set of structured questionnaires on parental mental health and HRQOL, parenting style, neighborhood cohesion, and their children's well-being and behaviors. Physical examination including blood pressure, heart rate, weight, height, and waist-to-hip ratio will also be carried out on both parents and children. A swab of buccal cells will be taken from each child. Venous blood will be sampled from each parent.

This study will have four assessment waves: Baseline, T2 follow up (6 months), T3 follow up (12 months), and T4 follow up (24 months). Physical health data and biological samples will be collected by research nurses and research assistants during health assessment session held in community centers. Questionnaire data will be collected by trained interviewers during telephone survey. To minimize attrition, a package of questionnaires and a sheet of instructions and equipment (i.e. brushes) for swab-taking at home may also be sent to parents upon request.

ELIGIBILITY:
Inclusion Criteria:

* Family monthly household income does not exceed 75% of Hong Kong's median monthly household income
* At least one parent and one child aged 6 to 16 years of the same family have given consent to participate in the main cohort study

Exclusion Criteria:

* Parents cannot speak or read Chinese;
* Children were born prematurely and/or with a congenital deformity; and
* Neither parent is the primary caregiver of the child.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants from low-income families will be recruited from the existing cohort study (main cohort study) on the effectiveness of the Trekkers Family Enhancement Scheme funded by a philanthropic foundation in Hong Kong (Kerry Group Kuok Foundation (Hong Kong) Limited).
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Child CHQ General Health Perception subscale score from baseline, 6 months, 12 months to 24 months | baseline, 6 months, 12 months and 24 months
  Quality of life: Child Health Questionnaire - Parent Form 50 (CHQ-PF50) is a parent proxy measure of children's physical and psychological wellbeing, with 50 items grouped into 12 multi-item subscales. Its Chinese version has been shown to have good psychometric properties in local Chinese children

SECONDARY OUTCOMES:
Change in Child SDQ Totally Difficulty score from baseline, 6 months, 12 months to 24 months | baseline, 6 months, 12 months and 24 months
  Strength and Difficulties Questionnaire (SDQ) is a 25-item parent-completed questionnaire measuring children's behavioral issues. The SDQ, with 5 subscales, has been translated into traditional Chinese and tested with satisfactory reliability and validity in local children.
Change in Child telomere length from baseline to 24 months | baseline and 24 months
  Telomere length will be measured by the method adapted from that originally published by Cawthon. For each sample, the telomere length will be represented by the relative ratio of the telomere repeat copy number (T) to the single copy gene 36BA copy number (S). The T/S ratio will be determined by quantitative polymerase chain reaction (qPcR) using a 7900HT Thermocycler (Applied Biosystems).
Change in Parental allostatic load index from baseline, 6 months, 12 months to 24 months | baseline, 12 months and 24 months
  A review of literature has identified a set of physiological parameters that can reflect allostatic load and yet be conveniently measured, including blood pressure, heart rate, body-mass-index, waist-to-hip ratio, lipid profile, fasting glucose and glycosylated haemoglobin. An index score of allostatic load will be calculated by summing the number of parameters that fall into the "highest" risk quartile defined by local clinical practice guidelines
Change in Parental SF-12v2 HRQOL scores from baseline, 6 months, 12 months to 24 months | baseline, 6 months, 12 months and 24 months
  The SF-12 Health Survey-Version 2 (SF-12v2) is a 12-item quality of life assessment instrument that covers 8 subscales. The Chinese version of SF-12v2 has been validated and normed in local Chinese population
Change in Parental DASS Stress subscale score from baseline, 6 months, 12 months to 24 months | baseline, 6 months, 12 months and 24 months
  Depression Anxiety Stress Scale (DASS) has 3 subscales, each with 7 items rating the severity/frequency of symptoms of stress, anxiety and depression respectively. DASS also has well-established psychometric properties and been validated in Chinese population.

OTHER OUTCOMES:
Parental PHQ-9-score, DASS Depression and Anxiety subscale score | 6 months
  Depression Anxiety Stress Scale (DASS) has 3 subscales, each with 7 items rating the severity/frequency of symptoms of stress, anxiety and depression respectively. DASS also has well-established psychometric properties and been validated in Chinese population. In addition, Patient Health Questionnaire - 9 (PHQ-9) will be used to screen for depression in parents. The Chinese version of PHQ-9 has been validated and used in previous local studies.
Family disharmony measured by FHS-5 | 6 months
  The Chinese version of Family Harmony Scale - 5 (FHS-5) will be used to measure family harmony.
Child physical assault and neglect potential measured by the Physical Assault and Neglect subscale of the CTSPC | 6 months
  Parental risk of physically abusing and neglecting children will also be assessed with the Child Physical Assault and Neglect subscale of the Parent Child Conflict Tactics Scale (CTSPC).
Authoritative parenting style measured by the Authoritative Parenting Style subscale of the PSDQ | 6 months
  Parenting style will be assessed using the Authoritative Parenting Style subscale of the Parenting Style and Dimension Questionnaire (PSDQ).
Neighbourhood cohesion measured by NCES | 6 months
  The Chinese version of Neighborhood Collective Efficacy Scale (NCES) is a 10-item scale, with five items each on informal social control and social cohesion.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yee Tak Yu, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong RSM, Yu EYT, Guo VY, Wan EY, Chin WY, Wong CKH, Fung CSC, Tung KTS, Wong WH, Ip P, Tiwari AFY, Lam CLK. A prospective cohort study to investigate parental stress and child health in low-income Chinese families: protocol paper. BMJ Open. 2018 Feb 22;8(2):e018792. doi: 10.1136/bmjopen-2017-018792. PMID 29472262